CLINICAL TRIAL: NCT02427620
Title: A Phase II Study of Ibrutinib Plus Rituximab With Hyper-CVAD Consolidation in Newly Diagnosed Young Patients With Mantle Cell Lymphoma: A Window Period for Bioimmunotherapy Before Chemotherapy
Brief Title: Ibrutinib, Rituximab, and Consolidation Chemotherapy in Treating Young Patients With Newly Diagnosed Mantle Cell Lymphoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-0559; NCI-2015-00960 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2014-0559 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2015-04-15; First posted 2015-04-28 (Estimated); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Blastoid Variant Mantle Cell Lymphoma; Mantle Cell Lymphoma; Pleomorphic Variant Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — Cyclophosphamide; Cytarabine; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Doxorubicin; ibrutinib; Methotrexate; merphos; Rituximab; CT-P10; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (ibrutinib, rituximab, consolidation chemotherapy) (Experimental): PART I (IBRUTINIB PLUS RITUXIMAB): Patients receive ibrutinib PO QD on days 1-28 and rituximab IV over 6-8 hours on days 1, 8, 15, and 22 of cycle 1 and then over 4 hours on day 1 of cycles 3-12. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity or until patients achieve complete response.
  PART II (CONSOLIDATION THERAPY): Patients receive rituximab IV over 6 hours on day 1; dexamethasone PO or IV on days 1-4; cyclophosphamide IV over 3 hours BID on days 2-4; doxorubicin hydrochloride IV over 15-30 minutes on day 5; and vincristine sulfate IV over 15-30 minutes on day 5 of cycles 1, 3, 5, and 7. Patients also receive rituximab IV over 6 hours on day 1; methotrexate IV over 24 hours on day 2; and cytarabine IV over 2 hours BID on days 3 and 4 of cycles 2, 4, 6, and 8. Treatment repeats every 28 days for up to 8 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Dexamethasone; Drug: Doxorubicin; Drug: Doxorubicin Hydrochloride; Drug: Ibrutinib; Other: Laboratory Biomarker Analysis; Drug: Methotrexate; Biological: Rituximab; Drug: Vincristine; Drug: Vincristine Sulfate

INTERVENTIONS:
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Dexamethasone — Given PO or IV
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Dxevo; Fluorodelta; Fortecortin; Gammacorten; Hemady; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
Drug: Doxorubicin — Given IV
  Other Names: Adriablastin; Hydroxydaunomycin; Hydroxyl Daunorubicin; Hydroxyldaunorubicin
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin HCl; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; hydroxydaunorubicin; Rubex
Drug: Ibrutinib — Given PO
  Other Names: BTK Inhibitor PCI-32765; CRA-032765; Imbruvica; PCI-32765
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Methotrexate — Given IV
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
Biological: Rituximab — Given IV
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Riabni; Rituxan; Rituximab ABBS; Rituximab ARRX; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar JHL1101; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; Rituximab Biosimilar SIBP-02; rituximab biosimilar TQB2303; Rituximab PVVR; rituximab-abbs; Rituximab-arrx; Rituximab-pvvr; RTXM83; Ruxience; Truxima
Drug: Vincristine — Given IV
  Other Names: Leurocristine; VCR; Vincrystine
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine Sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate

SUMMARY:
This phase II trial studies how well ibrutinib, rituximab, and consolidation chemotherapy consisting of cyclophosphamide, vincristine sulfate, doxorubicin hydrochloride, dexamethasone, methotrexate, and cytarabine work in treating young patients with newly diagnosed mantle cell lymphoma. Ibrutinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Immunotherapy with monoclonal antibodies, such as rituximab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Drugs used in chemotherapy, such as cyclophosphamide, vincristine sulfate, doxorubicin hydrochloride, dexamethasone, methotrexate, and cytarabine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving more than one drug (combination chemotherapy) may kill more cancer cells. Giving ibrutinib together with rituximab and consolidation chemotherapy may be a better treatment for mantle cell lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the response rate of ibrutinib plus rituximab in young newly diagnosed mantle cell lymphoma (MCL) including young high-risk patients.

SECONDARY OBJECTIVES:

I. To evaluate the progression free survival of ibrutinib plus rituximab with rituximab - cyclophosphamide, vincristine (vincristine sulfate), doxorubicin (doxorubicin hydrochloride), and dexamethasone (hyper-CVAD) consolidation in newly diagnosed MCL patients and in high-risk patients.

II. To further evaluate the toxicity profile of the ibrutinib/rituximab combination and consolidation therapy.

III. To estimate the rate of complete response (CR) prior to and following consolidation therapy.

IV. To estimate the response duration and overall survival. V. To analyze progression free survival in a subgroup of patients presenting with high risk features after receiving an additional 2 years of maintenance therapy with rituximab and ibrutinib at doses used in part 1 of the study, starting after part 2 of the study ends.

OUTLINE:

PART I (IBRUTINIB PLUS RITUXIMAB): Patients receive ibrutinib orally (PO) once daily (QD) on days 1-28 and rituximab intravenously (IV) over 6-8 hours on days 1, 8, 15, and 22 of cycle 1 and then over 4 hours on day 1 of cycles 3-12. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity or until patients achieve complete response.

PART II (CONSOLIDATION THERAPY): Patients receive rituximab IV over 6 hours on day 1; dexamethasone PO or IV on days 1-4; cyclophosphamide IV over 3 hours twice daily (BID) on days 2-4; doxorubicin hydrochloride IV over 15-30 minutes on day 5; and vincristine sulfate IV over 15-30 minutes on day 5 of cycles 1, 3, 5, and 7. Patients also receive rituximab IV over 6 hours on day 1; methotrexate IV over 24 hours on day 2; and cytarabine IV over 2 hours BID on days 3 and 4 of cycles 2, 4, 6, and 8. Treatment repeats every 28 days for up to 8 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 4 months for 2 years, every 6 months for 2 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patient has a confirmed diagnosis of mantle cell lymphoma with CD20 positivity in tissue biopsy
* Patients with MCL must be symptomatic and need immediate therapy; symptoms and nature of MCL include any of the following:

  * Blastoid variant
  * Pleomorphic variant
  * B symptoms
  * Mantle Cell International Prognostic Score (MIPI) > 3
  * Ki-67 >= 30%
  * Bulky tumors > 7 cm or in case of >= 2 tumors, each >= 5 cm in diameter
  * Disease threatening organ function
  * Elevated lactate dehydrogenase (LDH)
  * Peripheral blood white blood cell (PB WBC) > 50,000
  * Pancytopenia due to bone marrow MCL
  * Patient's choice due to anxiety
  * Pain due to lymphoma
  * Somatic mutations in the TP53, c-MYC or NOTCH genes
  * Size of spleen >= 20 cm
* Patients with mantle cell lymphoma with any of the following will be considered "high-risk" for the purpose of this protocol:

  * Blastoid or pleomorphic histology
  * Ki-67 index larger than 30%
  * Bulky tumor of larger than 7 cm or in case of multiple tumors, larger than or equal to 5 cm each in diameter
  * Somatic mutations in the TP53, c-MYC or NOTCH genes
  * Size of spleen >= 20 cm
* Patient has newly diagnosed disease with no prior therapy
* Understand and voluntarily sign an Institutional Review Board (IRB)-approved informed consent form
* Age =< 65 years at the time of signing the informed consent
* Patients should have bi-dimensional measurable disease using the Cheson criteria (measurable disease by computed tomography [CT] scan defined as at least 1 lesion that measures >= 1.5 cm in single dimension)
* Gastrointestinal or bone marrow or spleen only patients are allowable
* Eastern Cooperative Oncology Group (ECOG) performance status of 2 or less
* An absolute neutrophil count (ANC) > 1,000/mm^3 (patients who have bone marrow infiltration by MCL are eligible if their ANC is >= 500/mm^3 [growth factor allowed]; these patients should be discussed with either the principal investigator [PI] or Co-PI of the study for final approval)
* Platelet count > 100,000/mm^3 (patients who have bone marrow infiltration by MCL are eligible if their platelet level is equal to or > than 20,000/mm^3; these patients should be discussed with either the PI or Co-PI of the study for final approval)
* Serum bilirubin < 1.5 mg/dl
* Creatinine (Cr) clearance >= 30 mL/min
* Aspartate transaminase (AST)/serum glutamic oxaloacetic transaminase (SGOT) and alanine transaminase (ALT)/serum glutamic-pyruvate transaminase (SGPT) < 2 x upper limit of normal or < 5 x upper limit of normal if hepatic metastases are present; Gilbert's disease is allowed
* Cardiac ejection fraction >= 50% by echocardiogram (ECHO) or multiple gated acquisition scan (MUGA)
* Disease free of prior malignancies with exception of currently treated basal cell, squamous cell carcinoma of the skin, carcinoma "in situ" of the cervix or breast, or other malignancies in remission (including prostate cancer patients in remission from radiation therapy, surgery or brachytherapy), not actively being treated
* Females of childbearing potential (FCBP)* must have a negative serum or urine pregnancy test (within 30 days of initiation of protocol therapy) and must be willing to use acceptable methods of birth control; men must agree to use a latex condom during sexual contact with a female of childbearing potential even if they have had a successful vasectomy

  * A female of childbearing potential is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)

Exclusion Criteria:

* Any serious medical condition including but not limited to, uncontrolled hypertension, uncontrolled diabetes mellitus, active/symptomatic coronary artery disease, chronic obstructive pulmonary disease (COPD), renal failure, active hemorrhage, or psychiatric illness that, in the investigators opinion places the patient at unacceptable risk and would prevent the subject from signing the informed consent form
* Pregnant or breast feeding females
* Known human immunodeficiency virus (HIV) infection
* Patients with active hepatitis B or C infection (not including patients with prior hepatitis B vaccination); these patients should be cleared by gastrointestinal (GI) consultation for hepatitis B and infectious disease consult for hepatitis C
* All patients with central nervous system lymphoma
* Significant neuropathy (grades 3 - 4, or grade 2 with pain) within 14 days prior to enrollment
* Contraindication to any of the required concomitant drugs or supportive treatments or intolerance to hydration due to preexisting pulmonary or cardiac impairment including pleural effusion requiring thoracentesis or ascites requiring paracentesis unless due to lymphoma
* Malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel or ulcerative colitis, symptomatic inflammatory bowel disease, or partial or complete bowel obstruction, or any other gastrointestinal condition that could interfere with the absorption and metabolism of ibrutinib
* Major surgery within 4 weeks of initiation of therapy; clearance letter from primary physician required
* Requires anticoagulation with warfarin or equivalent vitamin K antagonist
* Requires treatment with strong cytochrome P4503A (CYP3A) inhibitors
* Patients with New York Heart Association (NYHA) class III and IV heart failure, myocardial infarction in the preceding 6 months, and significant conduction abnormalities, including but not limited to 2nd degree atrioventricular block (AV block) type II, 3rd degree block, QT prolongation (corrected QT [QTc] > 500 millisecond [msec]), sick sinus syndrome, ventricular tachycardia, symptomatic bradycardia (heart rate < 50 beats per minute [bpm]), hypotension, light headedness and syncope; patients with persistent and uncontrolled atrial fibrillation will be excluded; the protocol excludes patients who have recently had a stent and by recommendation of their cardiologist need to stay on anticoagulants such as warfarin or equivalent vitamin K antagonist
* Acute infection requiring treatment (IV antibiotics, antivirals, or antifungals) within 14 days prior to initiation of study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Estimated)
Dates: Start 2015-06-03 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (complete response + partial response) | At 8 weeks
  Will be monitored using the Bayesian stopping boundaries calculated based on beta-binomial distribution. Logistic regression will be utilized to assess the effect of patient prognostic factors on the response rate.

SECONDARY OUTCOMES:
Incidence of adverse events | At 4 weeks
  Will be monitored using the Bayesian stopping boundaries calculated based on beta-binomial distribution. Logistic regression will be utilized to assess the effect of patient prognostic factors on the toxicity rate. Toxicity data by type and severity will be summarized by frequency tables.
Overall survival | Up to 6 years
  Will be estimated using the method of Kaplan and Meier. Comparison of time-to-event endpoints by important subgroups will be made using the log-rank test.
Progression free survival | Up to 6 years
  Will be estimated using the method of Kaplan and Meier. Comparison of time-to-event endpoints by important subgroups will be made using the log-rank test.

CONTACTS AND LOCATIONS:
Overall Officials: Luhua (Michael) Wang, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Wang ML, Jain P, Zhao S, Lee HJ, Nastoupil L, Fayad L, Ok CY, Kanagal-Shamanna R, Hill HA, Yao Y, Hagemeister FB, Westin JR, Fowler N, Samaniego F, Steiner R, Nair R, Iyer SP, Navsaria L, Badillo M; Mantle Cell Research Group; Feng L, Xuelin H, Nogueras Gonzalez GM, Xu G, Wagner-Bartak N, Thirumurthi S, Santos D, Tang G, Lin P, Wang SA, Jorgensen J, Yin CC, Li S, Patel KP, Vega F, Medeiros LJ, Flowers CR, Wang L. Ibrutinib-rituximab followed by R-HCVAD as frontline treatment for young patients (</=65 years) with mantle cell lymphoma (WINDOW-1): a single-arm, phase 2 trial. Lancet Oncol. 2022 Mar;23(3):406-415. doi: 10.1016/S1470-2045(21)00638-0. Epub 2022 Jan 21. PMID 35074072
- [Derived] Jain P, Zhao S, Lee HJ, Hill HA, Ok CY, Kanagal-Shamanna R, Hagemeister FB, Fowler N, Fayad L, Yao Y, Liu Y, Moghrabi OB, Navsaria L, Feng L, Nogueras Gonzalez GM, Xu G, Thirumurthi S, Santos D, Iliescu C, Tang G, Medeiros LJ, Vega F, Avellaneda M, Badillo M, Flowers CR, Wang L, Wang ML. Ibrutinib With Rituximab in First-Line Treatment of Older Patients With Mantle Cell Lymphoma. J Clin Oncol. 2022 Jan 10;40(2):202-212. doi: 10.1200/JCO.21.01797. Epub 2021 Nov 19. PMID 34797699
- [Derived] Jain P, Romaguera J, Srour SA, Lee HJ, Hagemeister F, Westin J, Fayad L, Samaniego F, Badillo M, Zhang L, Nastoupil L, Kanagal-Shamanna R, Fowler N, Wang ML. Four-year follow-up of a single arm, phase II clinical trial of ibrutinib with rituximab (IR) in patients with relapsed/refractory mantle cell lymphoma (MCL). Br J Haematol. 2018 Aug;182(3):404-411. doi: 10.1111/bjh.15411. Epub 2018 May 22. PMID 29785709
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org